CLINICAL TRIAL: NCT01938846
Title: An Open Label Phase I Dose Finding Study of BI 860585 Administered Orally in a Continuous Dosing Schedule as Single Agent and in Combination With Exemestane or With Paclitaxel in Patients With Various Advanced and/or Metastatic Solid Tumours
Brief Title: BI 860585 Dose Escalation Single Agent and in Combination With Exemestane or With Paclitaxel in Patients With Various Advanced and/or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1325.1; 2013-000765-36 (EudraCT Number)
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — exemestane; Paclitaxel

ARMS (3):
- BI 860585 (Experimental): Multiple ascending doses of BI 860585 administered continuously in a 28-day cycle, including food interaction cohorts
  Interventions: Drug: BI 860585
- BI 860585 + paclitaxel (Experimental): Multiple ascending doses of BI 860585 in combination with fixed dose paclitaxel
  Interventions: Drug: BI 860585; Drug: paclitaxel
- BI 860585 + exemestane (Experimental): Multiple ascending doses of BI 860585 in combination with fixed dose exemestane
  Interventions: Drug: exemestane; Drug: BI 860585

INTERVENTIONS:
Drug: BI 860585 — BI 860585 multiple dose escalation, once daily
  Arms: BI 860585 + paclitaxel
Drug: exemestane — exemestane once daily
  Arms: BI 860585 + exemestane
Drug: BI 860585 — BI 860585 multiple dose escalation, once daily
  Arms: BI 860585
Drug: BI 860585 — BI 860585 multiple dose escalation, once daily
  Arms: BI 860585 + exemestane
Drug: paclitaxel — paclitaxel once weekly
  Arms: BI 860585 + paclitaxel

SUMMARY:
The primary objective of the trial is to determine the maximum tolerated doses (MTD) of BI 860585 alone and in combination with exemestane or paclitaxel. To determine the MTDs, patients are entered sequentially into escalating dose cohorts. Secondary objectives are objective response and disease control according to RECIST criteria version 1.1

ELIGIBILITY:
Inclusion criteria:

* Patients with histologically or cytologically confirmed diagnosis of advanced, measurable or evaluable, non-resectable and/or metastatic solid tumours, which has shown to be progressive;
* Patients who have received previous standard of care therapy for their disease and have progressed;
* 18 years or older;
* Life expectancy >= 3 months;
* Written informed consent in accordance with International Conference on Harmonisation/Good Clinical Practice (ICH/GCP) and local legislation;
* Eastern Cooperative Oncology Group (ECOG), performance score 0-2.

Additional inclusion criteria for the combination arms:

* Patients must have confirmed progressive disease within the last 6 months, (in case of measurable disease, progression should be confirmed according to Response Evaluation Criteria in Solid Tumours (RECIST) criteria version 1.1;
* Patients carrying a tumour for whom treatment with either exemestane or paclitaxel would be considered appropriate by the investigator;

Additional inclusion criteria for expansion part:

* Patients must have measurable progressive disease within the last 6 months documented/proven according to RECIST criteria version 1.1.
* Patients entering the expansion cohorts must also have:
* Arm A: any advanced/metastatic solid tumour suitable for biopsy and must have provided informed consent for biopsy and biomarker analysis.
* Arm B: any cytologically or histologically confirmed ER+ (estrogen receptor positive) advanced/metastatic solid tumours for which treatment with exemestane would be considered appropriate by the investigator.
* Arm C: any advanced/metastatic solid tumour for which treatment with paclitaxel would be considered appropriate by the investigator.

Exclusion criteria:

* Serious concomitant non-oncological disease/illness considered by the investigator to be incompatible with the protocol;
* Patients with untreated or symptomatic brain metastases;
* Second malignancies requiring active therapy;
* Clinical Congestive Heart Failure (CHF) Grade III-IV;
* Myocardial infarction within the last 6 months prior to inclusion, or symptomatic coronary artery disease;
* Adequate bone marrow, liver and renal function;
* Patients with known HIV/hepatitis/active infectious disease considered by the investigator to be incompatible with the protocol;
* Patients unable to take oral medication;
* Chronic diarrhoea or other gastrointestinal disorders;
* Treatment with anti-cancer-therapies: cytotoxic or standard chemotherapy, immunotherapy, radiotherapy, biological therapies, molecular targeted or other investigational drugs, within four weeks of the first treatment with the study medication (or within one week for non-cytotoxic drugs);
* Recovery from previous surgery and anticancer medical treatments;
* Hypersensitivity to combination drugs or excipients;
* Patients with a history of uncontrolled diabetes mellitus.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-09-05 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2017-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (4):
- Belgium (2):
  - Brussels - UNIV Saint-Luc, Brussels
  - UNIV UZ Gent, Ghent
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera di Parma, Parma

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label, Phase I, dose-finding study of BI 860585, a total of 90 patients received at least one dose of study medication.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites which would then ensure that all patients met all inclusion/exclusion criteria. Patients were not to be entered to trial treatment if any one of the specific entry criteria were not met.
Groups:
- BI 860585 Monotherapy: Patients were administered with BI 860585 daily oral dose of 5 milligram starting dose) over 28-day treatment courses
- BI 860585 + Exemestane: Patients were administered with daily oral dose of BI 860585 in combination with 25 milligram/day standard fixed dose of Exemestane over 28-day treatment courses
- BI 860585 + Paclitaxel: Patients were administered with BI 860585 in combination with Paclitaxel weekly intravenous infusion of 60 milligram/meter^2 for the first dose level/treatment cohort and 80 milligram/meter^2 (the standard combination dose) for subsequent dose levels/treatment cohorts over 28-day treatment courses
Period: Overall Study
Arm/Group | BI 860585 Monotherapy | BI 860585 + Exemestane | BI 860585 + Paclitaxel
Started (Entered/randomised) | 41 | 25 | 24
Completed (Not discontinued from last trial medication) | 0 | 0 | 0
Not Completed | 41 | 25 | 24
Not completed — Progressive disease | 26 | 18 | 16
Not completed — Adverse Event | 8 | 4 | 3
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Other than listed | 5 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set includes all patients who were administered at least one dose of any study medication (BI 860585, exemestane, or paclitaxel).
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 860585 Monotherapy | BI 860585 + Exemestane | BI 860585 + Paclitaxel | Total
Number analyzed (Participants) | 41 | 25 | 24 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of signing informed consent form is presented. Population: TS
  Years | 58.4 (13.8) | 58.3 (9.5) | 58.5 (10.2) | 58.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of subjects is categorized as Male or Female. Population: TS
  Participants
    Female | 13 | 23 | 12 | 48
    Male | 28 | 2 | 12 | 42

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Dose-Limiting Toxicities (DLTs) in the First Course of Each Treatment Arm
Description: The number of patients with Dose-Limiting Toxicities (DLTs) in the first course of each treatment arm to identify the Maximum Tolerated Dose (MTD) for BI 860585 monotherapy and BI 860585 in combination with exemestane of paclitaxel.
Time Frame: 28 days (Maximum tolerated dose (MTD) evaluation period (First Treatment Cycle))
Population: Treated and Evaluable Set: The treated and evaluable set includes all patients who were administered at least one dose of study medication and who are evaluable with respect to DLT in the MTD evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | BI 860585 Monotherapy | BI 860585 + Exemestane | BI 860585 + Paclitaxel
Number analyzed (Participants) | 36 | 21 | 18
Participants
  Total with dose limiting toxicities | 4 | 4 | 2

2. Primary Outcome: The Maximum Tolerated Dose (MTD) for Each Treatment Arm
Description: The Maximum Tolerated Dose (MTD) for each treatment arm was the dose that was 1 dose cohort below that at which ≥2 of 6 patients had experienced DLT. i.e., the MTD was the highest dose studied for which the DLT incidence was no more than 17% (i.e. 1 of 6 patients) during the first treatment course.
Time Frame: 28 days (Maximum tolerated dose (MTD) evaluation period (First Treatment Cycle))
Population: as for outcome 1
Measure: Number; unit: Milligram (mg)
Arm/Group | BI 860585 Monotherapy | BI 860585 + Exemestane | BI 860585 + Paclitaxel
Number analyzed (Participants) | 36 | 21 | 18
Milligram (mg)
  BI 860585 | 220 | 160 | 160
  Exemestane | NA — Not applicable for this arm | 25 | NA — Not applicable for this arm
  Paclitaxel | NA — Not applicable for this arm | NA — Not applicable for this arm | 80

3. Secondary Outcome: Objective Response Rate (Complete Response or Partial Response as Per the Response Evaluation Criteria In Solid Tumors Criteria [RECIST], Version 1.1)
Description: As Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for objective response rate (Complete Response (CR), disappearance of all target lesions; Partial Response (PR), =30% decrease in the sum of the longest diameter of target lesions) for target lesions assessed by Magnetic resonance imaging (MRI) and Computed tomography (CT)
Time Frame: From the date of first treatment administration until the earliest of disease progression, death, or last adequate tumour assessment before new anti-cancer therapy; data collected up to cut-off date 30 Jun 2017, Up to 1389 days
Population: Treated Set: The treated set includes all patients who were administered at least one dose of any study medication (BI 860585, exemestane or paclitaxel).
Measure: Count of Participants; unit: Participants
Arm/Group | BI 860585 Monotherapy | BI 860585 + Exemestane | BI 860585 + Paclitaxel
Number analyzed (Participants) | 41 | 25 | 24
Participants | 0 | 4 | 5

4. Secondary Outcome: Disease Control Rate/Clinical Benefit Rate (Complete Response, Partial Response or Stable Disease as Per Response Evaluation Criteria In Solid Tumors Criteria [RECIST], Version 1.1)
Description: As Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for disease control rate/clinical benefit rate (Complete Response (CR), disappearance of all target lesions; Partial Response (PR), =30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression) for target lesions assessed by Magnetic resonance imaging (MRI) and Computed tomography (CT)
Time Frame: From the date of first treatment administration until the earliest of disease progression, death, or last adequate tumour assessment before new anti-cancer therapy.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | BI 860585 Monotherapy | BI 860585 + Exemestane | BI 860585 + Paclitaxel
Number analyzed (Participants) | 41 | 25 | 24
Participants | 8 | 7 | 14

5. Secondary Outcome: Duration of Clinical Benefit
Description: Duration of clinical benefit (Disease control) was defined as the time between first treatment administration until the earliest of disease progression or death, for patients with disease control.
Time Frame: as for outcome 3
Population: Patients with disease control from the treated set (Treated Set: The treated set includes all patients who were administered at least one dose of any study medication (BI 860585, exemestane or paclitaxel)).
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | BI 860585 Monotherapy | BI 860585 + Exemestane | BI 860585 + Paclitaxel
Number analyzed (Participants) | 8 | 7 | 14
Months | 8.31 (4.78) | 10.06 (7.26) | 7.79 (3.30)

6. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response was defined as the time from first objective response until the earliest of progression or death, for patients with objective response.
Time Frame: as for outcome 3
Population: Patients with objective response from the treated set (Treated Set: The treated set includes all patients who were administered at least one dose of any study medication (BI 860585, exemestane or paclitaxel)).
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | BI 860585 Monotherapy | BI 860585 + Exemestane | BI 860585 + Paclitaxel
Number analyzed (Participants) | 0 | 4 | 5
Months |  | 9.16 (9.83) | 4.42 (3.06)

7. Secondary Outcome: Area Under the Concentration-time Curve in Plasma of BI 860585 Over the Time Interval From 0 to Infinity (AUC0-∞)
Description: AUC0-∞, area under the concentration-time curve in plasma of BI 860585 over the time interval from 0 to infinity after single administration of BI 860585
Time Frame: Pharmacokinetic samples were collected at pre-dose and 0.5, 1, 2, 3, 4, 6, 8 and 23.917 hours after administration of BI 860585.
Population: Pharmacokinetic Analysis Set (PKS): This patient set includes all evaluable patients in the treated set (TS) which provide at least one observation for at least one pharmacokinetic (PK) endpoint without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol*hour/ Litre [nmol*h/L]
Groups:
- 5 mg BI 860585: Continuous daily oral dose of 5 milligram/day (starting dose) over 28-day treatment courses of BI 860585 Monotherapy
- 10 mg BI 860585: Continuous daily oral dose of 10 milligram/day over 28-days treatment courses of BI 860585 Monotherapy
- 20 mg BI 860585: Continuous daily oral dose of 20 milligram/day over 28-days treatment courses of BI 860585 Monotherapy
- 40 mg BI 860585: Continuous daily oral dose of 40 milligram/day over 28-days treatment courses of BI 860585 Monotherapy
- 80 mg BI 860585: Continuous daily oral dose of 80 milligram/day over 28-days treatment courses of BI 860585 Monotherapy
- 120 mg BI 860585: Continuous daily oral dose of 120 milligram/day over 28-days treatment courses of BI 860585 Monotherapy
- 160 mg BI 860585: Continuous daily oral dose of 160 milligram/day over 28-days treatment courses of BI 860585 Monotherapy
- 220 mg BI 860585: Continuous daily oral dose of 220 milligram/day over 28-days treatment courses of BI 860585 Monotherapy
- 300 mg BI 860585: Continuous daily oral dose of 300 milligram/day over 28-days treatment courses of BI 860585 Monotherapy
- 40 mg BI 860585+25 mg Exemestane: Continuous daily oral dose of 25 mg/day standard fixed dose of exemestane over 28-day treatment courses combination with 40 mg BI 860585
- 80 mg BI 860585+25 mg Exemestane: Continuous daily oral dose of 25 mg/day standard fixed dose of exemestane over 28-day treatment courses combination with 80 mg BI 860585
- 120 mg BI 860585+25 mg Exemestane: Continuous daily oral dose of 25 mg/day standard fixed dose of exemestane over 28-day treatment courses combination with 120 mg BI 860585
- 160 mg BI 860585+25 mg Exemestane: Continuous daily oral dose of 25 mg/day standard fixed dose of exemestane over 28-day treatment courses combination with 160 mg BI 860585
- 80 mg BI 860585+60 mg/m^2 Paclitaxel: Patients were administered with 80 mg BI 860585 in combination with weekly intravenous infusion of 60 mg/m^2 the standard combination dose of paclitaxel for the first dose level/treatment for subsequent dose levels/treatment cohorts over 28-day treatment courses
- 80 mg BI 860585+80 mg/m^2 Paclitaxel: Patients were administered with 80 mg BI 860585 in combination with weekly intravenous infusion of 80 mg/m^2 the standard combination dose of paclitaxel for the first dose level/treatment for subsequent dose levels/treatment cohorts over 28-day treatment courses
- 120 mg BI 860585+80 mg/m^2 Paclitaxel: Patients were administered with 120 mg BI 860585 in combination with weekly intravenous infusion of 80 mg/m^2 the standard combination dose of paclitaxel for the first dose level/treatment for subsequent dose levels/treatment cohorts over 28-day treatment courses
- 160 mg BI 860585+80 mg/m^2 Paclita: Continuous daily oral dose of 160 mg BI 860585 in combination with once weekly iv infusion of 80 mg/m^2 paclitaxel
Arm/Group | 5 mg BI 860585 | 10 mg BI 860585 | 20 mg BI 860585 | 40 mg BI 860585 | 80 mg BI 860585 | 120 mg BI 860585 | 160 mg BI 860585 | 220 mg BI 860585 | 300 mg BI 860585 | 40 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+25 mg Exemestane | 120 mg BI 860585+25 mg Exemestane | 160 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+60 mg/m^2 Paclitaxel | 80 mg BI 860585+80 mg/m^2 Paclitaxel | 120 mg BI 860585+80 mg/m^2 Paclitaxel | 160 mg BI 860585+80 mg/m^2 Paclita
Number analyzed (Participants) | 3 | 2 | 2 | 3 | 3 | 0 | 5 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
nanomol*hour/ Litre [nmol*h/L] | 21100 (27.3) | 51100 (65.4) | 70300 (26.4) | 126000 (17.7) | 425000 (28.5) |  | 680000 (38.9) | 791000 (12.3) | 1030000 (10.5) |  |  |  |  |  |  |  |

8. Secondary Outcome: Area Under the Concentration-time Curve in Plasma of BI 860585 Over the Time Interval From 0 to 24 Hours (AUC0-24)
Description: AUC0-24, area under the concentration-time curve in plasma of BI 860585 over the time interval from 0 to 24 hours after single administration of BI 860585
Time Frame: as for outcome 7
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol*hour/ Litre [nmol*h/L]
Arm/Group | 5 mg BI 860585 | 10 mg BI 860585 | 20 mg BI 860585 | 40 mg BI 860585 | 80 mg BI 860585 | 120 mg BI 860585 | 160 mg BI 860585 | 220 mg BI 860585 | 300 mg BI 860585 | 40 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+25 mg Exemestane | 120 mg BI 860585+25 mg Exemestane | 160 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+60 mg/m^2 Paclitaxel | 80 mg BI 860585+80 mg/m^2 Paclitaxel | 120 mg BI 860585+80 mg/m^2 Paclitaxel | 160 mg BI 860585+80 mg/m^2 Paclita
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 3 | 5 | 5 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
nanomol*hour/ Litre [nmol*h/L] | 12900 (20.0) | 23400 (30.7) | 45400 (29.6) | 83200 (24.7) | 236000 (15.6) | 299000 (21.1) | 401000 (21.4) | 470000 (6.09) | 641000 (8.43) |  |  |  |  |  |  |  |

9. Secondary Outcome: Half Life of BI 860585 (t1/2)
Description: t ½, half-life of BI 860585 in plasma over a dosing interval after single administration of BI 860585
Time Frame: as for outcome 7
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour (h)
Arm/Group | 5 mg BI 860585 | 10 mg BI 860585 | 20 mg BI 860585 | 40 mg BI 860585 | 80 mg BI 860585 | 120 mg BI 860585 | 160 mg BI 860585 | 220 mg BI 860585 | 300 mg BI 860585 | 40 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+25 mg Exemestane | 120 mg BI 860585+25 mg Exemestane | 160 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+60 mg/m^2 Paclitaxel | 80 mg BI 860585+80 mg/m^2 Paclitaxel | 120 mg BI 860585+80 mg/m^2 Paclitaxel | 160 mg BI 860585+80 mg/m^2 Paclita
Number analyzed (Participants) | 3 | 2 | 2 | 3 | 3 | 0 | 5 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hour (h) | 17.1 (14.5) | 21.6 (50.1) | 15.6 (11.8) | 14.2 (27.2) | 19.7 (28.0) |  | 17.2 (33.7) | 17.4 (11.0) | 16.9 (6.14) |  |  |  |  |  |  |  |

10. Secondary Outcome: Maximum Measured Concentration of BI 860585 (Cmax)
Description: Cmax, maximum measured concentration of BI 860585 in plasma over a dosing interval after single administration of BI 860585
Time Frame: as for outcome 7
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Litre [nmol/L]
Arm/Group | 5 mg BI 860585 | 10 mg BI 860585 | 20 mg BI 860585 | 40 mg BI 860585 | 80 mg BI 860585 | 120 mg BI 860585 | 160 mg BI 860585 | 220 mg BI 860585 | 300 mg BI 860585 | 40 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+25 mg Exemestane | 120 mg BI 860585+25 mg Exemestane | 160 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+60 mg/m^2 Paclitaxel | 80 mg BI 860585+80 mg/m^2 Paclitaxel | 120 mg BI 860585+80 mg/m^2 Paclitaxel | 160 mg BI 860585+80 mg/m^2 Paclita
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
nanomole/Litre [nmol/L] | 995 (26.3) | 1590 (21.5) | 3330 (4.76) | 6770 (37.6) | 16900 (15.0) | 18800 (16.4) | 28000 (36.0) | 32400 (18.5) | 51500 (10.7) |  |  |  |  |  |  |  |

11. Secondary Outcome: Time to Maximum Concentration of BI 860585 (Tmax)
Description: Tmax, Time to maximum concentration of BI 860585 in plasma over a dosing interval after single administration of BI 860585
Time Frame: as for outcome 7
Population: PKS
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | 5 mg BI 860585 | 10 mg BI 860585 | 20 mg BI 860585 | 40 mg BI 860585 | 80 mg BI 860585 | 120 mg BI 860585 | 160 mg BI 860585 | 220 mg BI 860585 | 300 mg BI 860585 | 40 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+25 mg Exemestane | 120 mg BI 860585+25 mg Exemestane | 160 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+60 mg/m^2 Paclitaxel | 80 mg BI 860585+80 mg/m^2 Paclitaxel | 120 mg BI 860585+80 mg/m^2 Paclitaxel | 160 mg BI 860585+80 mg/m^2 Paclita
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hour (h) | 3.03 [1.98 to 3.03] | 4.00 [2.00 to 8.00] | 3.00 [1.07 to 3.17] | 2.00 [1.00 to 5.98] | 3.00 [1.05 to 3.00] | 6.00 [3.00 to 8.02] | 3.47 [2.00 to 8.00] | 3.00 [2.00 to 6.00] | 2.00 [2.00 to 3.20] |  |  |  |  |  |  |  |

12. Secondary Outcome: Area Under the Concentration-time Curve of BI 860585 in Plasma Over a Dosing Interval at Steady State (AUCτ,ss)
Description: AUCτ,ss, area under the concentration-time curve of BI 860585 in plasma over the dosing interval at steady state after multiple administration of BI 860585 (Day 22) in BI 860585 monotherapy and in combination with exemestane and paclitaxel.
Time Frame: Pharmacokinetic samples were collected at pre-dose and at 504.5, 505, 506, 507, 508, 510, 512, 527.917 hours after drug administration.
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol*hour/ Litre [nmol*h/L]
Arm/Group | 5 mg BI 860585 | 10 mg BI 860585 | 20 mg BI 860585 | 40 mg BI 860585 | 80 mg BI 860585 | 120 mg BI 860585 | 160 mg BI 860585 | 220 mg BI 860585 | 300 mg BI 860585 | 40 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+25 mg Exemestane | 120 mg BI 860585+25 mg Exemestane | 160 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+60 mg/m^2 Paclitaxel | 80 mg BI 860585+80 mg/m^2 Paclitaxel | 120 mg BI 860585+80 mg/m^2 Paclitaxel | 160 mg BI 860585+80 mg/m^2 Paclita
Number analyzed (Participants) | 3 | 2 | 2 | 3 | 3 | 0 | 5 | 5 | 3 | 3 | 3 | 5 | 7 | 2 | 0 | 4 | 3
nanomol*hour/ Litre [nmol*h/L] | 32000 (9.28) | 63100 (86.1) | 103000 (3.91) | 163000 (6.34) | 442000 (21.8) |  | 840000 (23.9) | 838000 (24.3) | 1350000 (12.3) | 271000 (12.9) | 281000 (31.8) | 676000 (30.7) | 988000 (19.1) | 374000 (4.69) |  | 630000 (54.8) | 730000 (20.3)

13. Secondary Outcome: Half Life of BI 860585 at Steady State (t1/2,ss)
Description: t1/2,ss, half-life of BI 860585 in plasma at steady state after multiple administration of BI 860585 (Day 22) in BI 860585 monotherapy and in combination with exemestane and paclitaxel.
Time Frame: as for outcome 12
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour (h)
Arm/Group | 5 mg BI 860585 | 10 mg BI 860585 | 20 mg BI 860585 | 40 mg BI 860585 | 80 mg BI 860585 | 120 mg BI 860585 | 160 mg BI 860585 | 220 mg BI 860585 | 300 mg BI 860585 | 40 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+25 mg Exemestane | 120 mg BI 860585+25 mg Exemestane | 160 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+60 mg/m^2 Paclitaxel | 80 mg BI 860585+80 mg/m^2 Paclitaxel | 120 mg BI 860585+80 mg/m^2 Paclitaxel | 160 mg BI 860585+80 mg/m^2 Paclita
Number analyzed (Participants) | 3 | 2 | 2 | 3 | 3 | 0 | 5 | 5 | 0 | 3 | 3 | 5 | 7 | 0 | 0 | 4 | 0
Hour (h) | 31.5 (8.73) | 28.9 (47.4) | 33.1 (10.2) | 21.3 (20.0) | 29.8 (7.67) |  | 27.6 (18.3) | 24.9 (22.2) |  | 22.9 (13.8) | 24.7 (68.4) | 23.3 (7.82) | 25.3 (25.9) |  |  | 24.2 (37.2) |

14. Secondary Outcome: Time to Maximum Concentration of BI 860585 at Steady State (Tmax,ss)
Description: tmax,ss, Time to maximum concentration of BI 860585 at steady state after multiple administration of BI 860585 (Day 22) in BI 860585 monotherapy and in combination with exemestane and paclitaxel.
Time Frame: as for outcome 12
Population: PKS
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | 5 mg BI 860585 | 10 mg BI 860585 | 20 mg BI 860585 | 40 mg BI 860585 | 80 mg BI 860585 | 120 mg BI 860585 | 160 mg BI 860585 | 220 mg BI 860585 | 300 mg BI 860585 | 40 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+25 mg Exemestane | 120 mg BI 860585+25 mg Exemestane | 160 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+60 mg/m^2 Paclitaxel | 80 mg BI 860585+80 mg/m^2 Paclitaxel | 120 mg BI 860585+80 mg/m^2 Paclitaxel | 160 mg BI 860585+80 mg/m^2 Paclita
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 5 | 5 | 2 | 3 | 3 | 5 | 7 | 2 | 4 | 4 | 4
Hour (h) | 6.00 [1.95 to 6.00] | 2.02 [2.02 to 4.00] | 2.00 [1.00 to 4.07] | 3.00 [2.02 to 3.18] | 2.00 [0.983 to 3.03] | 3.61 [3.00 to 7.97] | 3.10 [2.98 to 4.05] | 3.03 [2.08 to 6.00] | 5.00 [2.00 to 8.00] | 3.98 [2.00 to 4.00] | 2.00 [1.00 to 2.97] | 3.00 [1.00 to 6.00] | 2.02 [1.50 to 4.02] | 2.03 [2.00 to 2.05] | 4.92 [3.05 to 8.12] | 2.50 [1.00 to 3.00] | 6.00 [3.98 to 8.00]

15. Secondary Outcome: Maximum Measured Concentration of BI 860585 in Plasma at Steady State (Cmax,ss)
Description: Cmax,ss, maximum measured concentration at steady state after multiple administration of BI 860585 (Day 22) in BI 860585 monotherapy and in combination with exemestane and paclitaxel.
Time Frame: as for outcome 12
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol/ Litre [nmol/L]
Arm/Group | 5 mg BI 860585 | 10 mg BI 860585 | 20 mg BI 860585 | 40 mg BI 860585 | 80 mg BI 860585 | 120 mg BI 860585 | 160 mg BI 860585 | 220 mg BI 860585 | 300 mg BI 860585 | 40 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+25 mg Exemestane | 120 mg BI 860585+25 mg Exemestane | 160 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+60 mg/m^2 Paclitaxel | 80 mg BI 860585+80 mg/m^2 Paclitaxel | 120 mg BI 860585+80 mg/m^2 Paclitaxel | 160 mg BI 860585+80 mg/m^2 Paclita
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 5 | 5 | 2 | 3 | 3 | 5 | 7 | 2 | 4 | 4 | 4
nanomol/ Litre [nmol/L] | 1730 (18.5) | 3720 (47) | 6630 (0.832) | 11600 (21.5) | 29700 (28.2) | 33700 (26.6) | 50100 (16.7) | 50500 (27.1) | 75700 (17.5) | 16700 (3.63) | 19600 (31.2) | 43800 (30.5) | 61400 (25.7) | 20500 (13.8) | 20700 (39.6) | 38900 (56.4) | 35400 (40.7)

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after last drug administration; up to 209 weeks
Description: The treated set (includes all patients who were administered at least one dose of any study medication (BI 860585, exemestane, or paclitaxel)) was used for safety analysis.
Groups:
- 40 mg BI 860585+25 mg Exemestane: Patients were administered with daily oral dose of 40 mg BI 860585 in combination with 25 mg exemestane standard fixed dose over 28-day treatment courses
- 80 mg BI 860585+25 mg Exemestane: Patients were administered with daily oral dose of 80 mg BI 860585 in combination with 25 mg exemestane standard fixed dose over 28-day treatment courses
- 120 mg BI 860585+25 mg Exemestane: Patients were administered with daily oral dose of 120 mg BI 860585 in combination with 25 mg exemestane standard fixed dose over 28-day treatment courses
- 160 mg BI 860585+25 mg Exemestane: Patients were administered with daily oral dose of 160 mg BI 860585 in combination with 25 mg exemestane standard fixed dose over 28-day treatment courses
- 220 mg BI 860585+25 mg Exemestane: Patients were administered with daily oral dose of 220 mg BI 860585 in combination with 25 mg exemestane standard fixed dose over 28-day treatment courses
- 160 mg BI 860585+80 mg/m^2 Paclitaxel: Patients were administered with 160 mg BI 860585 in combination with weekly intravenous infusion of 80 mg/m^2 the standard combination dose of paclitaxel for the first dose level/treatment for subsequent dose levels/treatment cohorts over 28-day treatment courses
- 220 mg BI 860585+80 mg/m^2 Paclitaxel: Patients were administered with 220 mg BI 860585 in combination with weekly intravenous infusion of 80 mg/m^2 the standard combination dose of paclitaxel for the first dose level/treatment for subsequent dose levels/treatment cohorts over 28-day treatment courses
Arm/Group | 5 mg BI 860585 | 10 mg BI 860585 | 20 mg BI 860585 | 40 mg BI 860585 | 80 mg BI 860585 | 120 mg BI 860585 | 160 mg BI 860585 | 220 mg BI 860585 | 300 mg BI 860585 | 40 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+25 mg Exemestane | 120 mg BI 860585+25 mg Exemestane | 160 mg BI 860585+25 mg Exemestane | 220 mg BI 860585+25 mg Exemestane | 80 mg BI 860585+60 mg/m^2 Paclitaxel | 80 mg BI 860585+80 mg/m^2 Paclitaxel | 120 mg BI 860585+80 mg/m^2 Paclitaxel | 160 mg BI 860585+80 mg/m^2 Paclitaxel | 220 mg BI 860585+80 mg/m^2 Paclitaxel
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 1/3 | 0/3 | 0/3 | 1/7 | 1/7 | 0/9 | 0/3 | 0/3 | 3/4 | 1/7 | 0/8 | 0/3 | 0/3 | 0/4 | 0/7 | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 2/3 | 1/3 | 2/3 | 4/7 | 4/7 | 4/9 | 2/3 | 0/3 | 4/4 | 3/7 | 2/8 | 1/3 | 2/3 | 3/4 | 3/7 | 4/7 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 7/7 | 7/7 | 9/9 | 3/3 | 3/3 | 4/4 | 7/7 | 8/8 | 3/3 | 3/3 | 4/4 | 7/7 | 7/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5 mg BI 860585 (N=3) | 10 mg BI 860585 (N=3) | 20 mg BI 860585 (N=3) | 40 mg BI 860585 (N=3) | 80 mg BI 860585 (N=3) | 120 mg BI 860585 (N=7) | 160 mg BI 860585 (N=7) | 220 mg BI 860585 (N=9) | 300 mg BI 860585 (N=3) | 40 mg BI 860585+25 mg Exemestane (N=3) | 80 mg BI 860585+25 mg Exemestane (N=4) | 120 mg BI 860585+25 mg Exemestane (N=7) | 160 mg BI 860585+25 mg Exemestane (N=8) | 220 mg BI 860585+25 mg Exemestane (N=3) | 80 mg BI 860585+60 mg/m^2 Paclitaxel (N=3) | 80 mg BI 860585+80 mg/m^2 Paclitaxel (N=4) | 120 mg BI 860585+80 mg/m^2 Paclitaxel (N=7) | 160 mg BI 860585+80 mg/m^2 Paclitaxel (N=7) | 220 mg BI 860585+80 mg/m^2 Paclitaxel (N=3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Condition aggravated (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perihepatic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral oesophagitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaesthetic complication pulmonary (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neurological decompensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aorto-duodenal fistula (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5 mg BI 860585 (N=3) | 10 mg BI 860585 (N=3) | 20 mg BI 860585 (N=3) | 40 mg BI 860585 (N=3) | 80 mg BI 860585 (N=3) | 120 mg BI 860585 (N=7) | 160 mg BI 860585 (N=7) | 220 mg BI 860585 (N=9) | 300 mg BI 860585 (N=3) | 40 mg BI 860585+25 mg Exemestane (N=3) | 80 mg BI 860585+25 mg Exemestane (N=4) | 120 mg BI 860585+25 mg Exemestane (N=7) | 160 mg BI 860585+25 mg Exemestane (N=8) | 220 mg BI 860585+25 mg Exemestane (N=3) | 80 mg BI 860585+60 mg/m^2 Paclitaxel (N=3) | 80 mg BI 860585+80 mg/m^2 Paclitaxel (N=4) | 120 mg BI 860585+80 mg/m^2 Paclitaxel (N=7) | 160 mg BI 860585+80 mg/m^2 Paclitaxel (N=7) | 220 mg BI 860585+80 mg/m^2 Paclitaxel (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 2 | 2 | 2 | 1 | 2 | 3 | 3 | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Maculopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 2 | 0 | 2 | 3 | 4 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 1 | 3 | 3 | 6 | 3 | 1 | 0 | 3 | 6 | 2 | 1 | 3 | 4 | 5 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 1 | 2 | 1 | 1 | 2 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 1 | 3 | 4 | 4 | 2 | 0 | 3 | 4 | 2 | 1 | 2 | 2 | 3 | 2 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0 | 3 | 2 | 0 | 2 | 0 | 0 | 3 | 5 | 2 | 2 | 1 | 1 | 2 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 0 | 4 | 3 | 4 | 1 | 0 | 3 | 3 | 0 | 1 | 1 | 1 | 2 | 1 | 1
Asthenia (General disorders) | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 2 | 1 | 2 | 1 | 2 | 5 | 3 | 2 | 2 | 3 | 4 | 2 | 2 | 3 | 5 | 6 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperpyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 2 | 2 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral oesophagitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 1
Ammonia increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 2 | 1 | 2 | 3 | 0 | 1 | 1 | 0 | 1 | 2
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 2 | 1 | 1 | 3 | 1 | 0 | 1 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 2 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 1 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 2 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 3 | 2 | 1 | 3 | 3 | 3 | 2 | 1 | 2 | 1 | 4 | 1 | 1 | 2 | 6 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 2 | 5 | 5 | 5 | 3 | 0 | 0 | 3 | 5 | 1 | 3 | 4 | 7 | 6 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 1 | 1 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 2 | 3 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head titubation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 3 | 0
Postural tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vesical fistula (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 0 | 2 | 3 | 0 | 1 | 1 | 1 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 3 | 3 | 2 | 0 | 0 | 3 | 3 | 2 | 0 | 1 | 3 | 2 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The trial was discontinued at the end of the dose-escalation phase for each treatment arm, before starting the expansion phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-08-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT01938846/SAP_000.pdf
  • Study Protocol (2015-02-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT01938846/Prot_001.pdf